CLINICAL TRIAL: NCT01738256
Title: Applicability and Efficiency of Different Approaches in Lifestyle Interventions - Lifestyle Management and Changes in Everyday Life
Brief Title: Study of Effectiveness of Different Lifestyle Interventions for Health and Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: SalWe Ltd. (Industry); University of Eastern Finland (Other); University of Helsinki (Other); VTT Technical Research Centre of Finland (Other); Finnish Institute of Occupational Health (Other); Finnish Red Cross Blood Service (Other); Duodecim Medical Publications Ltd. (Industry); Firstbeat Technologies Ltd. (Industry); Vivago Ltd (Unknown); Valio Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Salwe_27819_WP303.2-1
Record Dates: First submitted 2012-08-17; First posted 2012-11-30 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Metabolic Syndrome Risk Factors; Overweight; Psychological Stress
Keywords: Cognitive Behavior Therapy; Acceptance Commitment Therapy; Psychological Stress; Metabolic Syndrome; Overweight; Life Style
MeSH Terms: conditions — Overweight; Stress, Psychological; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Face-to-Face (Experimental): Group meetings face-to-face using intervention for wellbeing with ACT principles.
  Interventions: Behavioral: Wellbeing intervention (ACT)
- Mobile (Experimental): Intervention for wellbeing via mobile phone application with ACT principles.
  Interventions: Behavioral: Wellbeing intervention (ACT)
- Internet (Experimental): Intervention for wellbeing via Internet (Virtual Health Check and Coaching).
  Interventions: Behavioral: Wellbeing intervention (Internet)
- Control (Experimental): Control group, no intervention.
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: Wellbeing intervention (ACT) — The intervention is based on principles of acceptance-commitment therapy (ACT). It aims to increase psychological flexibility through different exercises that are developed for improving skills of being present, dealing with thoughts and feelings, as well as support clarifying individual values and value-based actions. In addition exercises for relaxation, physical activity, and mindful eating are provided. The content of intervention for face-to-face and mobile groups is similar but delivery method is different.
  Arms: Face-to-Face; Mobile
Behavioral: Wellbeing intervention (Internet) — The intervention is Duodecim Virtual Health Check and Coaching where the subject gets feedback based on his/her health information and is provided with different weekly tasks regarding lifestyle changes. The tasks are developed based on principles of cognitive behaviour therapy (CBT).
  Arms: Internet
Behavioral: No intervention — No intervention
  Arms: Control

SUMMARY:
The purpose of this study is to examine the effectiveness and applicability of different interventions designed for enhancing overall wellbeing. Lifestyle changes, as well as psychological and physiological health variables are assessed. The interventions are based on the principles of cognitive behavioural therapy, and delivered either face-to-face, via mobile phone application, or Internet.

DETAILED DESCRIPTION:
The study focuses on targeting overweight, stress, and impaired overall wellbeing with new cost-effective intervention methods. The intervention methods are based on the principles of cognitive behavioural therapy (CBT) and further acceptance-commitment therapy (ACT). The interventions are delivered either face-to-face, via mobile application, or via Internet. The purpose of each intervention is to improve the subjects lifestyles and activate them towards beneficial changes in their everyday life. The psychological and physiological effects of interventions are measured with various invasive and non-invasive methods. The study gives new insight into effectiveness and acceptability of up-to-date psychological intervention methods, and new knowledge of different ways to deliver interventions for improving wellbeing of an individual.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 27-34.9
* Psychological Stress (3/4 or 4/4 points in General Health Questionnaire)
* Possibility to use computer and internet connection

Exclusion Criteria:

* Diagnosed severe chronic illness

  * Symptomatic cardiovascular disease
  * Type 1 or 2 diabetes
  * Severe psychiatric conditions
  * Remarkable clinical operation within past 6 months
  * Heart attack or stroke within past 6 months
  * Kidney disease requiring Dialysis
* Regular use of cortisone pills
* Eating disorder: bulimia
* Disability pension for psychological reasons
* Pregnancy or breastfeeding within the pas 6 months
* Shift work (in three shifts) or night work
* Participation in other intervention studies during the present study

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 339 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Psychological Flexibility (AAQ-2) | Change from Baseline in Psychological Flexibility at 8.5 months

SECONDARY OUTCOMES:
Diet (interview, questionnaire) | pre, post, follow-up (0, 10, 36 weeks)
Perceived and physiological stress (questionnaire, heart rate variability measurement) | pre, post, follow-up (0, 10, 36 weeks)
Blood lipids | pre, post, follow-up (0, 10, 36)
Sleep (ESS, Basic Nordic Sleep Questionnaire, actigraphy, sleep diary) | pre, post, follow-up (0, 10, 36 weeks)
Physical Activity (questionnaire) | pre, post, follow-up (0, 10, 36 weeks)
User experiences concerning technology (interview, questionnaire) | during, post, follow-up (2, 10, 36 weeks)
Depression | Pre, post, follow-up (0, 10, 36 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Raimo Lappalainen, PhD, Principal Investigator — University of Jyvaskyla; Marjukka Kolehmainen, PhD, Principal Investigator — University of Eastern Finland; Miikka Ermes, PhD, Principal Investigator — VTT Technical Research Centre of Finland
Locations (3):
- Finland (3):
  - Institute of Biomedicine, University of Helsinki, Helsinki
  - Department of Psychology and Department of Health Sciences, University of Jyvaskyla, Jyväskylä
  - Institute of Public Health and Clinical Nutrition, University of Eastern Finland (UEF), Kuopio

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Jarvela-Reijonen E, Jarvinen S, Karhunen L, Fohr T, Myllymaki T, Sairanen E, Lindroos S, Peuhkuri K, Hallikainen M, Pihlajamaki J, Puttonen S, Korpela R, Ermes M, Lappalainen R, Kujala UM, Kolehmainen M, Laitinen J. Sleep-time physiological recovery is associated with eating habits in distressed working-age Finns with overweight: secondary analysis of a randomised controlled trial. J Occup Med Toxicol. 2021 Jun 28;16(1):23. doi: 10.1186/s12995-021-00310-6. PMID 34183032
- [Derived] Jarvela-Reijonen E, Puttonen S, Karhunen L, Sairanen E, Laitinen J, Kolehmainen M, Pihlajamaki J, Kujala UM, Korpela R, Ermes M, Lappalainen R, Kolehmainen M. The Effects of Acceptance and Commitment Therapy (ACT) Intervention on Inflammation and Stress Biomarkers: a Randomized Controlled Trial. Int J Behav Med. 2020 Oct;27(5):539-555. doi: 10.1007/s12529-020-09891-8. PMID 32394219
- [Derived] Jarvela-Reijonen E, Karhunen L, Sairanen E, Muotka J, Lindroos S, Laitinen J, Puttonen S, Peuhkuri K, Hallikainen M, Pihlajamaki J, Korpela R, Ermes M, Lappalainen R, Kolehmainen M. The effects of acceptance and commitment therapy on eating behavior and diet delivered through face-to-face contact and a mobile app: a randomized controlled trial. Int J Behav Nutr Phys Act. 2018 Feb 27;15(1):22. doi: 10.1186/s12966-018-0654-8. PMID 29482636
- [Derived] Mattila E, Lappalainen R, Valkkynen P, Sairanen E, Lappalainen P, Karhunen L, Peuhkuri K, Korpela R, Kolehmainen M, Ermes M. Usage and Dose Response of a Mobile Acceptance and Commitment Therapy App: Secondary Analysis of the Intervention Arm of a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2016 Jul 28;4(3):e90. doi: 10.2196/mhealth.5241. PMID 27468653
- [Derived] Lappalainen R, Sairanen E, Jarvela E, Rantala S, Korpela R, Puttonen S, Kujala UM, Myllymaki T, Peuhkuri K, Mattila E, Kaipainen K, Ahtinen A, Karhunen L, Pihlajamaki J, Jarnefelt H, Laitinen J, Kutinlahti E, Saarelma O, Ermes M, Kolehmainen M. The effectiveness and applicability of different lifestyle interventions for enhancing wellbeing: the study design for a randomized controlled trial for persons with metabolic syndrome risk factors and psychological distress. BMC Public Health. 2014 Apr 4;14:310. doi: 10.1186/1471-2458-14-310. PMID 24708617